CLINICAL TRIAL: NCT00532883
Title: Effectiveness of Hydroxyurea and Magnesium Pidolate Alone and in Combination in Hemoglobin SC Disease: A Phase II Trial
Brief Title: Hydroxyurea and Magnesium Pidolate to Treat People With Hemoglobin Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment has been terminated due to a slow rate of enrollment.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHAMPS-St. Jude; U54HL070587 (NIH)
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Hemoglobin SC Disease
Keywords: Sickle Cell Disease; Vaso-occlusive Event; Painful Crises; Acute Chest Syndrome
MeSH Terms: conditions — Hemoglobin SC Disease; Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome | interventions — Hydroxyurea; Pyrrolidonecarboxylic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Pills and Placebo Liquid (Placebo Comparator)
  Interventions: Other: Placebo Pills and Placebo Liquid
- Hydroxyurea Pills and Placebo Liquid (Active Comparator)
  Interventions: Drug: Hydroxyurea
- Placebo Pills and Magnesium Pidolate Liquid (Active Comparator)
  Interventions: Drug: Magnesium Pidolate
- Hydroxyurea Pills and Magnesium Pidolate Liquid (Active Comparator)
  Interventions: Drug: Hydroxyurea; Drug: Magnesium Pidolate

INTERVENTIONS:
Drug: Hydroxyurea — HU capsules (20 mg/kg/day for 11 months) Mg/Placebo liquid (0.6 mEq/kg/day for 11 months)
  Arms: Hydroxyurea Pills and Magnesium Pidolate Liquid; Hydroxyurea Pills and Placebo Liquid
Drug: Magnesium Pidolate — HU/Placebo capsules (20 mg/kg/day for 11 months) Mg liquid (0.6 mEq/kg/day for 11 months)
  Arms: Hydroxyurea Pills and Magnesium Pidolate Liquid; Placebo Pills and Magnesium Pidolate Liquid
Other: Placebo Pills and Placebo Liquid — HU/Placebo capsules (20 mg/kg/day for 11 months) Mg/Placebo liquid (0.6 mEq/kg/day for 11 months)
  Arms: Placebo Pills and Placebo Liquid

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause intense pain episodes. Hemoglobin SCD (HbSC) is a form of SCD that is characterized by dense red blood cells. The purpose of this study is to evaluate the safety and effectiveness of hydroxyurea and magnesium pidolate, alone and combined, at reducing red blood cell density and the frequency of pain episodes in people with HbSC.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." SCD is caused by an abnormal type of hemoglobin, which is a protein inside red blood cells that carries oxygen. HbSC is a form of SCD that is characterized by the presence of dense red blood cells. People with HbSC usually develop less severe SCD symptoms than people with the more common form of the disease. There are limited treatment approaches aimed specifically at modifying the abnormal state of red blood cells. Also, few combination therapy treatments have been studied. The medication hydroxyurea is currently used to prevent sickle cell crises and to decrease the need for blood transfusions. The dietary supplement magnesium has not been widely studied as a treatment for SCD, but it may prevent dehydration, which may decrease the frequency of sickle cell crises. The purpose of this study is to evaluate the safety and effectiveness of hydroxyurea and magnesium pidolate, alone and combined, at reducing red blood cell density and the frequency of sickle cell crises in people with HbSC.

This 1-year study will enroll people with HbSC. Participants will be randomly assigned to one of the following four treatment groups:

* Group 1 participants will receive placebo pills and placebo liquid.
* Group 2 participants will receive hydroxyurea pills and placebo liquid.
* Group 3 participants will receive placebo pills and magnesium pidolate liquid.
* Group 4 participants will receive hydroxyurea pills and magnesium pidolate liquid.

Participants will receive the hydroxyurea or placebo pills once a day and the magnesium pidolate or placebo liquid twice a day for 11 months. Study visits will occur every 2 weeks during the first 2 months of the study, once a month for the following 9 months, and then at Year 1. At each visit, a physical exam and blood collection will occur. Selected visits will also include urine collection and a pregnancy test for female participants. Throughout the study, participants will record their study medication use in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HbSC disease
* Hemoglobin level between 8 and 12.5 g/dL
* At least one vaso-occlusive event (e.g., pain, acute chest syndrome) in the 12 months prior to study entry. An episode of pain is defined as the occurrence of pain in the extremities, back, abdomen, chest, or head that lasts at least 2 hours; requires a visit to a hospital, emergency room, clinic, or provider's office; and is not explained except by SCD. Acute chest syndrome is defined as a new pulmonary infiltrate on a chest x-ray associated with a fever (greater than 38.5° C), tachypnea, wheezing, cough, or chest pain.
* Regular compliance with comprehensive care
* In a steady disease state and not experiencing an acute complication of SCD (i.e., no hospitalization, pain event, or episode of acute chest syndrome within the 1 month prior to study entry)

Exclusion Criteria:

* Previous transfusion with remaining hemoglobin A greater than 10%
* Previous treatment with hydroxyurea within the last 3 months
* Previous treatment with magnesium within the 3 months prior to study entry (including vitamins containing magnesium)
* Poor compliance with previous treatment regimens
* Liver dysfunction (SGPT greater than twice the upper limit of normal) within the 1 month prior to study entry
* Kidney dysfunction (creatinine greater than or equal to 1.0 mg/dL for participants less than 18 years of age; greater than or equal to 1.2 mg/dL for participants 18 years of age or older) within the 1 month prior to study entry
* Pregnant
* Ten or more hospital admissions for pain in the 12 months prior to study entry
* Daily use of narcotics
* Treatment with any investigational drug in the 3 months prior to study entry
* Less than 3% red blood cells with density greater than 41 g/dL (as measured by the ADVIA 120 system)
* Positive HIV test
* Other long-term illness or disorder other than SCD that could adversely affect performance in the study (e.g., tuberculosis)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winfred C. Wang, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital and Research Center, Oakland, California
  - University of California Davis, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Saint Christopher's Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Wang W, Brugnara C, Snyder C, Wynn L, Rogers Z, Kalinyak K, Brown C, Qureshi A, Bigelow C, Neumayr L, Smith-Whitley K, Chui DH, Delahunty M, Woolson R, Steinberg M, Telen M, Kesler K. The effects of hydroxycarbamide and magnesium on haemoglobin SC disease: results of the multi-centre CHAMPS trial. Br J Haematol. 2011 Mar;152(6):771-6. doi: 10.1111/j.1365-2141.2010.08523.x. Epub 2011 Jan 31. PMID 21275961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from October 2006 through June 2008 at 10 sites across the United States. Subjects were recruited from sickle cell specific clinics.
Pre-assignment Details: Subjects were screened to ensure specific laboratory measurement levels after enrollment but prior to randomization.
Groups:
- Hydroxyurea/Magnesium: Hydroxyurea (20 mg/kg/day) combined with liquid magnesium pidolate (0.6 mEq/kg/day).
- Hydroxyurea/Mg Placebo: Hydroxyurea (20 mg/kg/day) combined with liquid Mg placebo.
- HU Placebo/Magnesium: HU placebo combined with liquid magnesium pidolate (0.6 mEq/kg/day).
- HU Placebo/Mg Placebo: Placebo for both hydroxyurea (20 mg/kg/day) and liquid magnesium pidolate (0.6 mEq/kg/day).
Period: Overall Study
Arm/Group | Hydroxyurea/Magnesium | Hydroxyurea/Mg Placebo | HU Placebo/Magnesium | HU Placebo/Mg Placebo
Started | 11 | 12 | 10 | 11
Completed | 5 (Study terminated early.) | 5 (Study terminated early.) | 6 (Study terminated early.) | 6 (Study terminated early.)
Not Completed | 6 | 7 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Subject was Nonadherent | 0 | 1 | 1 | 0
Not completed — Early Study Termination | 4 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxyurea/Magnesium | Hydroxyurea/Mg Placebo | HU Placebo/Magnesium | HU Placebo/Mg Placebo | Total
Number analyzed (Participants) | 11 | 12 | 10 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 9 | 9 | 37
  Between 18 and 65 years | 1 | 3 | 1 | 2 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.5 (4.41) | 16.8 (12.6) | 14.8 (8.45) | 17.3 (12.41) | 16.7 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 3 | 4 | 19
  Male | 7 | 4 | 7 | 7 | 25
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 10 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Distribution of the Density of Hemoglobin SC Red Cells
Description: An individuals' percentage of red blood cells with density greater than 41 g/dL as measured by Advia.
Time Frame: measured 2 months after initiation of treatment
Population: ITT: All randomized subjects who receive any clinical trial material. Subjects in the ITT population will be classified according to the treatment group to which they were randomized, regardless of what study drug they received.
Measure: Mean (Standard Deviation); unit: percent of cells
Arm/Group | Hydroxyurea/Magnesium | Hydroxyurea/Mg Placebo | HU Placebo/Magnesium | HU Placebo/Mg Placebo
Number analyzed (Participants) | 11 | 12 | 10 | 11
percent of cells | 12.09 (5.075) | 11.16 (7.296) | 10.49 (4.572) | 12.79 (3.739)
Statistical Analysis 1: Comparison: Hydroxyurea/Magnesium vs Hydroxyurea/Mg Placebo vs HU Placebo/Magnesium vs HU Placebo/Mg Placebo; F-test from a longitudinal mixed model (controlling for baseline measurement)testing the hypothesis of no difference in mean percent dense cells between the four treatment groups at Visit 6. The study was originally powered to detect a difference of 20%, but it was stopped early; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis — This is a global test comparing all four treatment arms

ADVERSE EVENTS:
Groups:
- Hydroxyurea/Magnesium Pidolate: 20 mg/kg/day
- Hydroxyurea/Placebo: 0.6 mEq/kg/day
- Placebo/Magnesium Pidolate: 20 mg/kg/day HU + 0.6 mEq/kg/day Mg
Arm/Group | Hydroxyurea/Magnesium Pidolate | Hydroxyurea/Placebo | Placebo/Magnesium Pidolate | Placebo/Placebo
Serious Adverse Events (participants affected / at risk) | 3/11 | 2/12 | 3/10 | 2/11
Other Adverse Events (participants affected / at risk) | 9/11 | 10/12 | 9/10 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea/Magnesium Pidolate (N=11) | Hydroxyurea/Placebo (N=12) | Placebo/Magnesium Pidolate (N=10) | Placebo/Placebo (N=11)
Acute chest syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 3 (5) | 1 (3) | 3 (4) | 2 (3)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea/Magnesium Pidolate (N=11) | Hydroxyurea/Placebo (N=12) | Placebo/Magnesium Pidolate (N=10) | Placebo/Placebo (N=11)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (2) | 0 (0) | 2 (3)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial bruit (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (10) | 5 (6) | 1 (1) | 3 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myringitis bullous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral soft tissue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 6 (39) | 6 (18) | 4 (7) | 8 (32)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spleen palpable (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 2 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (2) | 3 (4) | 3 (4)

LIMITATIONS AND CAVEATS:
This study was stopped early due to slow enrollment. It should therefore be viewed as a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No